CLINICAL TRIAL: NCT05464342
Title: Integral Physiological Adaptations to Carbohydrate Periodization
Acronym: IPACP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: University of Nicosia (Other); University of Cyprus (Other)
Responsible Party: Principal Investigator, Giorgos K. Sakkas, Associate Professor, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EEBK/EΠ/2018/10
Record Dates: First submitted 2022-07-04; First posted 2022-07-19 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Sleepiness; Fatigue; Feeding Patterns; Daytime Sleepiness, Excessive
Keywords: sleep; Carbohydrate periodization; Dietary Intervention; Sports Nutrition; Chrononutrition; Chronobiology; Gut Microbiome; miRNA
MeSH Terms: conditions — Sleepiness; Fatigue; Feeding Behavior; Disorders of Excessive Somnolence

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial. The study is composed of three groups, differentiating on evening carbohydrate quantity and quality (glycaemic index) intake. The trial period will last for 1 month for all groups. Intervention includes lifestyle changes, targeting exercise, and diet. The design is parallel.
Who Masked: Outcomes Assessor
Masking Description: Parameters such as questionnaires' scores, polysomnography outcomes, indices of health, gut microbiome, miRNA and other data will be masked and coded for blind analysis by the main investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Evening LGI Carbohydrate Consumption (Experimental): Dietary Intervention: Consumption of Low Glyceamic Index (LGI) carbohydrates intake post-workout/evening.
  Interventions: Behavioral: Evening LGI Carbohydrate Consumption Group
- Evening HGI Carbohydrate Consumption (Experimental): Dietary Intervention: Consumption of High Glyceamic Index (HGI) carbohydrates intake post-workout/evening.
  Interventions: Behavioral: Evening HGI Carbohydrate Consumption
- Evening NO-CHO Carbohydrate Consumption (Experimental): Dietary Intervention: No consumption of carbohydrates intake post-workout/evening.
  Interventions: Behavioral: Evening NO-CHO Carbohydrate Consumption

INTERVENTIONS:
Behavioral: Evening LGI Carbohydrate Consumption Group — Participants will receive in the evening food with low glycemic index
  Arms: Evening LGI Carbohydrate Consumption
Behavioral: Evening HGI Carbohydrate Consumption — Participants will receive in the evening food with high glycemic index
  Arms: Evening HGI Carbohydrate Consumption
Behavioral: Evening NO-CHO Carbohydrate Consumption — Participants will receive in the evening a meal with no carbohydrates at all.
  Arms: Evening NO-CHO Carbohydrate Consumption

SUMMARY:
The purpose of this study is to examine the effect of long-term carbohydrate periodization protocols on sleep architecture, sleep quality, daytime sleepiness, physical performance, body composition, gut microbiome, and miRNA in healthy trained individuals.

DETAILED DESCRIPTION:
Athletic populations have been particularly susceptible to sleep inadequacies, experience several sleep issues, and fall below the age-specific sleep recommendations. However, it is well demonstrated that exercise does not impair sleep by itself, and furthermore, acute post-exercise nutrition could elevate the exercise-induced sleep-optimizing effect, with further benefits for the next physical performance. In line with these findings, in a metanalysis of clinical trials, it was shown that pre-bed carbohydrate availability resulted in significant alterations in sleep architecture. It is of utmost importance to highlight that throughout this metanalysis, it was revealed that no long-term nutrition intervention for sleep optimization has been studied yet. These data raise the question of whether a long-term carbohydrate periodization protocol could optimize sleep and alter gut function in a way that athletic performance will be also enhanced. This would allow elucidating further potential interrelations and biological pathways underlying these adaptations.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes, Age between 18 and 50 yrs old, Regularly participating in sports activities.

Exclusion Criteria:

* Any kind of history of major diseases or medication, Excessive amounts of alcohol and caffeine consumption

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Sleep Efficiency | Assessed at 0-month (pre) and at 1-month (post)
  Changes sleep efficiency assessed by the gold-standard method of polysomnography. Sleep efficiency is the percentage of time spent asleep while in bed. It is calculated by dividing the amount of time spent asleep (in minutes) by the total amount of time in bed (in minutes). A normal sleep efficiency is considered to be 85% or higher.
Quality of Sleep Score | Assessed at 0-month (pre) and at 1-month (post)
  Changes in Quality of Sleep will be assessed by the Pittsburgh Sleep Quality Index. The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as the global score) indicating worse sleep quality.
Daytime Sleepiness | Assessed at 0-month (pre) and at 1-month (post)
  Changes in Daytime sleepiness will be assessed by Epworth Sleepiness Scale (ESS). The Epworth Sleepiness Scale (ESS) measures the general level of daytime sleepiness. It is a subjective scale that asks the respondent to rate his or her propensity to doze or fall asleep during 8 common daily activities to determine the level of daytime sleepiness. The score varies between 0-24 with 0-5 Lower Normal Daytime Sleepiness, 6-10 Higher Normal Daytime Sleepiness, 11-12 Mild Excessive Daytime Sleepiness, 13-15 Moderate Excessive Daytime Sleepiness, 16-24 Severe Excessive Daytime Sleepiness.

SECONDARY OUTCOMES:
Body Composition | Assessed at 0-month (pre) and at 1-month (post)
  Changes in Body composition. The changes in body composition will be assessed by the skinfold measurements and BIA
Exercise Performance | Assessed at 0-month (pre) and at 1-month (post)
  Changes in Exercise Performance will be assessed by a VO2max test. A VO2 max test is a maximal exercise test performed on a treadmill or bike while connected to a machine capable of analyzing your expired air. Your test provides data on how much oxygen you use as you exercise and determines the maximal oxygen you can consume during exercise.
Gut Microbiome | Assessed at 0-month (pre) and at 1-month (post)
  Changes in Gut Microbiome. Participants' gut microbiome will be studied by analyzing stool samples DNA will be extracted, and the presence of selected gut bacterial populations will be examined qualitatively and quantitatively using specific primers and quantitative Real-Time PCR.
miRNA levels | Assessed at 0-month (pre) and at 1-month (post)
  Changes in miRNA levels. miRNA levels that are associated with hypertrophy or cardiovascular function will be analyzed by blood sample collection at baseline and at one month.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Sakkas, PhD, Study Chair — University of Thessaly
Locations (2):
- Department of Life and Health Sciences, Nicosia, Cyprus
- Lifestlye Medicine Laboratory, TEFAA, University of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vlahoyiannis A, Andreou E, Aphamis G, Felekkis K, Pieri M, Sakkas GK, Giannaki CD. Evaluating the evening carbohydrate dilemma: the effect of within-the-day carbohydrate periodization on body composition and physical fitness. Eur J Nutr. 2024 Nov 25;64(1):23. doi: 10.1007/s00394-024-03540-6. PMID 39585451
- [Derived] Vlahoyiannis A, Andreou E, Bargiotas P, Aphamis G, Sakkas GK, Giannaki CD. The effect of chrono-nutritional manipulation of carbohydrate intake on sleep macrostructure: A randomized controlled trial. Clin Nutr. 2024 Mar;43(3):858-868. doi: 10.1016/j.clnu.2024.02.016. Epub 2024 Feb 15. PMID 38367595